CLINICAL TRIAL: NCT00750165
Title: Auto CPAP Based Energy Spectrum Analysis of Flow for Treatment of Obstructive Sleep Apnea Hypopnea Syndrome.
Brief Title: Auto Continuous Positive Airway Pressure (CPAP) Based Energy Spectrum Analysis of Flow for Treatment of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSA CPAP; 254 Validation, NYU
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Humidification; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Titration Night (Experimental): Treatment with the Fisher & Paykel Sleep Style 200 Auto CPAP device
  Interventions: Device: SleepStyle 200 Auto Series CPAP Humidifier

INTERVENTIONS:
Device: SleepStyle 200 Auto Series CPAP Humidifier — The device is a standard CPAP machine with a built in computer controller that incorporates software for evaluation of the flow signal obtained from the CPAP machine
  Other Names: HC254

SUMMARY:
Nasal Continuous Positive Airway Pressure (CPAP) is the standard therapy for obstructive sleep apnea hypopnea syndrome (OSAHS). This is most commonly administered as a single positive pressure that has been individualized for the patient to prevent obstructive respiratory events. However, the therapeutic pressure may vary by sleep stage and body position within a single night and may change over the course of several nights. One approach to dealing with this variability is the use of automatically adjusting CPAP that responds to patient breathing patterns with alterations in the delivered pressure. This study is designed to determine the effectiveness of using the energy spectrum analysis of flow signals to automatically adjust CPAP pressure and improve sleep variables. Thirty subjects who require CPAP will be recruited from the NYU sleep disorders center. Following diagnostic studies (either split night or full night) the subject will undergo a night of treatment with the Fisher and Paykel Healthcare AutoPAP. Efficacy of treatment will be evaluated based on normalization of sleep disordered breathing while treated with the AutoPAP.

ELIGIBILITY:
Inclusion Criteria:

* AHI >15 on the diagnostic portion of the study
* >18 years of age

Exclusion Criteria:

* Significant Central Apnea
* Congestive Heart Failure
* Inability to give informed consent
* Patient intolerance to CPAP
* Anatomical or physiological conditions making CPAP therapy inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Rapoport, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Sleep Disorders Center, New York, New York, United States

REFERENCES:
- [Background] Norman RG, Rapoport DM, Ayappa I. Detection of flow limitation in obstructive sleep apnea with an artificial neural network. Physiol Meas. 2007 Sep;28(9):1089-100. doi: 10.1088/0967-3334/28/9/010. Epub 2007 Sep 5. PMID 17827656
- See also: Sponsor website — http://fphcare.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Titration Night
Started | 32
Completed | 21
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Titration Night
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 51 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: The Apnea Hypopnea Index (AHI) measure of severity of Obstructive Sleep Apnea (OSA). It is a calculation of the number of apnea events and the number of hypopnea events divided by the total sleep time. Mild OSA is characterized between 5-15 events per hour. Moderate OSA is characterized as 15-30 events per hour. Severe OSA is characterized as greater than 30 events per hour.
Time Frame: 1 night
Measure: Mean (Full Range); unit: events per hour
Arm/Group | Titration Night
Number analyzed (Participants) | 21
events per hour | 2.4 [0.0 to 8.6]

2. Secondary Outcome: Percent of Time With Less Than 90% Oxygen Saturation
Description: Oxygen saturation is a measurement of the amount of oxygen present in the blood. An oxygen saturation of less than 90% is considered low, resulting in hypoxemia. Normal blood oxygen level is considered between 95-100%.
Time Frame: 1 Night
Measure: Mean (Full Range); unit: percentage of total sleep time
Arm/Group | Titration Night
Number analyzed (Participants) | 21
percentage of total sleep time | 1.4 [0 to 24.7]

3. Secondary Outcome: Respiratory Disturbance Index (RDI)
Description: Similar to AHI, the RDI is a calculation of the total number of respiratory disturbances in sleep. The calculation includes apneas and hypopneas, but also includes respiratory effort related arousals.
Time Frame: 1 Night
Measure: Mean (Full Range); unit: events per hour
Arm/Group | Titration Night
Number analyzed (Participants) | 21
events per hour | 7.1 [1.5 to 13.2]

4. Secondary Outcome: Arousal Index (AI)
Description: The Arousal Index is a calculation of the frequency of awakenings per hour of sleep. The higher the number, the more awakenings per hour.
Time Frame: 1 Night
Measure: Mean (Full Range); unit: events per hour
Arm/Group | Titration Night
Number analyzed (Participants) | 21
events per hour | 16.2 [4.9 to 32.9]

ADVERSE EVENTS:
Time Frame: 1 night
Arm/Group | Titration Night
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 6/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration Night (N=21)
Mask Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Difficulty Exhaling Due to Pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disruption of Sleep Due to Lab Environment (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No